CLINICAL TRIAL: NCT05898737
Title: The Interest of the Nociception Index (Nociception Level Index, NOL Index) for the Evaluation of Obstetric Pain Under Epidural Analgesia: a Prospective Pilot Study
Brief Title: Nociception Level Index (NOL Index) for Obstetrical Pain Assessment Under Epidural Analgesia.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: B0762023230305
Record Dates: First submitted 2023-04-17; First posted 2023-06-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Labor Pain; Nociceptive Pain; Epidural Analgesia; NOL Index
Keywords: Labor pain; Epidural analgesia; NOL Index
MeSH Terms: conditions — Labor Pain; Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturients: Parturients on labour requiring an epidural
  Interventions: Device: NOL-Index

INTERVENTIONS:
Device: NOL-Index — NOL Index monitoring with the PMD100™ (Medasense Biometrics Ltd.)
  Other Names: PMD100™ (Medasense Biometrics Ltd., Ramat Yishai, Israel)

SUMMARY:
Pain has been defined by the International Association for the Study of Pain (IASP) as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage". Labour pain is the pain experienced during labour and childbirth and it's characterised by nociceptive pain accompanied by sympathetic activation.

Since more than fifty years, the development of hospital obstetric assistance for labour, allowed the implementation of the pain relief culture in the demanding parturients population.

The ideal labour analgesic technique should provide consistent pain relief at any stage of labour, have a long duration of action, while being safe both for the mother and the foetus. It should also anticipate undesirable side effects, such as motor block.

The current gold standard for obstetric analgesia is the lumbar epidural technique using the administration of local anesthetics combined with opioids. However, the best administration mode is currently under debate, the main interest being the local anesthetic sparing responsible for various maternal side effects and the quality of maternal analgesia.

Despite the intense research in the field, the evaluation of the labour pain remains difficult as performed by the midwife and the anesthesiologist based on the patient's behaviour and her subjective self-assessment.

The PMD100™ (Medasense Biometrics Ltd., Ramat Yishai, Israel) is a non-invasive multiparametric nociception monitoring that has proved its interest in the intraoperative evaluation of patient's physiological response to pain under general anesthesia, using the NOL index variation. Nonetheless, it has been barely investigated in patients receiving locoregional anesthesia and never in the context of obstetrical pain.

The investigators support the idea that the NOL index monitoring could allow us to assess the degree of nociceptive stimulation related to obstetric labour and its variation under epidural analgesia, as well as to compare the efficacy of sensitive block using different epidural administration modes.

The aim of this pilot study is to evaluate the NOL Index variation during labour pain management with epidural analgesia.

The investigators will focus on the evaluation of analgesia in relation with the self-reported pain intensity, and secondly, the characteristics of the sensory block, the hemodynamic variables and side effects.

DETAILED DESCRIPTION:
1. Design:

   The investigators will conduct a prospective, repeated measures, monocentric, observational pilot study.

   The study will be carried out in the anesthesia department of the Saint Pierre University Hospital in collaboration with the obstetrics department.

   Parturient women in labour admitted into the delivery room, during the beginning of the first stage of labour demanding for an epidural will be recruited after signed written informed consent.

   The number of patients to be included has been calculated to be 55.
2. Anesthetic management:

   An epidural will be placed, initiated and maintained by the investigators according to the department's usual practice (including monitoring, technique and pump protocol).

   The epidural will be considered successful when the sensitive block has reached a T10 level within maximum 30 minutes.

   If the patient is not relieved within 30 minutes a new bolus readministration will be administered by the Patient-Controlled Epidural Analgesia (PCEA) pump.

   In case of:
   * Dura mater breach : exclusion of the patient from the protocol
   * Venous puncture : epidural replacement at another level
   * Hypotension (defined as a 20% drop in baseline blood pressure) needing vasopressors
   * Hypotension and fetal heart rate abnormalities
3. Nociception monitoring NOL Index is based on several variables nonlinear combination of heart rate, heart rate variability, photoplethysmograph wave amplitude, skin conductance, skin conductance fluctuations, and their time derivatives and variation upon activation of the sympathetic nervous system in response to a stimuli. The normal range of the NOL index has been set between 10 and 25, a value above 25 indicates that the patient is experiencing a nociceptive stimulation.

The monitoring will be placed on the contralateral side to the non invasive blood pressure (NIBP) upon recruitment and it will be calibrated during 30 seconds to 2 minutes period of time without uterine contraction, objectified by the toco monitoring and confirmed by the parturient before epidural placement.

Consented patients will be taught how to use the 0-10 numeric rating scales (NRS) to report pain intensity (where zero indicates no pain and 10 indicates the worst possible pain).

The NOL monitor will be hidden throughout the procedure, to reduce any bias during self-reporting.

The patient will be asked to report the self-evaluated pain at each contraction using the NRS scale during the initial 15 minutes following the initial bolus.

The characteristics of the block achieved (sensory and motor), analgesic and hemodynamic variables will be collected throughout the study period (1 hour after the implementation of the epidural) at several time points as follows :

T0 - Epidural request T1 - End of loading dose (bolus) T2 - Loading dose + 15 mins T3 - Loading dose + 30 mins T4 - Loading dose + 45 mins T5 - Loading dose + 60 mins

If a supplementary bolus is needed (PCEA) all the aforementioned variables will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old, able to self-report
* American Society of Anesthesiologists (ASA) score I to II
* Gestational age > 36 weeks of amenorrhea
* Primiparous or multiparous
* In labour
* Request and indication for epidural analgesia
* Height 160-175cm
* Intensity of pain objectified by Visual Analogue Scale (VAS) > 3/10

Exclusion Criteria:

* Patient refusal
* Contraindications to epidural analgesia (allergy to local anesthetics, coagulopathy, local infections)
* BMI > 40 kg/m2
* Weight > 110kg
* History of caesarean section
* Pre-eclampsia or pregnancy-induced hypertension
* Cardiac arrhythmias (including atrial fibrillation)
* Treatment with β-blockers
* Chronic opioid use
* History of substance abuse/dependency
* Psychiatric pathology (including depression, psychosis, etc.)
* Total language barrier
* Epidurals at uncomfortable times (night)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Parturient population
Study Population: Pregnant women in labour requesting an epidural analgesia
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
NOL Index variation (Delta-NOL) | 1 hour after the epidural implementation
  NOL Index variation between nociceptive (contraction) and non-nociceptive (rest) periods following the implementation of the epidural

SECONDARY OUTCOMES:
Nociception level | 1 hour after the epidural implementation
  Mesured by the NOL Index value (0-100). Higher scores meaning higher nociceptive stimuli.
Parturient's self-reported pain intensity | 1 hour after the epidural implementation
  Numerical Rating Scale (NRS) by the patient (0-10). Higher scores meaning more painful stimuli.
Maternal satisfaction | 1 hour after the epidural implementation
  Yes/no answer
Sensory block | 1 hour after the epidural implementation
  Sensory block using the cold ether test (maximal anatomical dermatome with a sensory block).
Motor block | 1 hour after the epidural implementation
  Motor block using the modified Bromage scale (0-4). Higher scores meaning more motor block.
Local anesthetic total dose | 1 hour after the epidural implementation
  Total dose of local anesthetics received by the epidural (mg)
Opioids total dose | 1 hour after the epidural implementation
  Total dose of opioids received by the epidural (mcg)
Need for PCEA rescue bolus | 1 hour after the epidural implementation
  Number of supplementary boluses if patient is unconfortable after 20 minutes.
Need of change in pump parameters | 1 hour after the epidural implementation
  Number of changes in pump parameters if patient is unconfortable after 20 minutes.
Blood pressure | 1 hour after the epidural implementation
  Systolic and diastolic blood pressure, measured by the non invasive blood pressure cuff (mmHg)
Heart rate | 1 hour after the epidural implementation
  Mesured by pulse oximetry (bpm)
Oxygen saturation | 1 hour after the epidural implementation
  Mesured by pulse oximetry (%)
Symptomatic hypotension | 1 hour after the epidural implementation
  Side effects such as symptomatic hypotension (yes/no answer).
Nausea/vomiting | 1 hour after the epidural implementation
  Side effects such as nausea/vomiting (yes/no answer).

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, MD, PhD, Study Director — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- CHU Saint-Pierre, Brussels, Bruxelles-Capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No